CLINICAL TRIAL: NCT00432939
Title: Primary Hyperparathyroidism: Non-classical Manifestations
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Shonni J. Silverberg, Professor of Medicine, Endocrinology, Columbia University
Other Study IDs: AAAB1955; R01DK066329 (NIH)
Record Dates: First submitted 2007-02-06; First posted 2007-02-08 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Primary Hyperparathyroidism
Keywords: Primary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Specimens of frozen serum will be retained for possible future analyses.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a research study to investigate cardiovascular health in people with mild hyperparathyroidism. Previous research has suggested that severe hyperparathyroidism may be associated with abnormalities in the heart and blood vessels. It is unclear whether mild hyperparathyroidism affects cardiovascular health. This study involves the investigation of the heart and blood vessels of people with mild hyperparathyroidism. Various non-invasive laboratory and radiological test to assess cardiovascular and bone health will be done at set intervals over the course of 2 years. It is our hypothesis that patients with primary hyperparathyroidism will have subtle abnormalities in their cardiovascular system. Using state-of-the art techniques that are sufficiently sensitive to detect these subtle abnormalities, we will define cardiovascular features of this disease that have, up to now, eluded clear definition. We expect taht the extent of these findings will be related to the severity of the underlying primary hyperparathyroidism. We further hypothesize that cardiovascular manifestations may regress with successful cure of the hyperparathyroid state.

DETAILED DESCRIPTION:
This study involves a total of 4 visits over a 2-year period. A variety of tests to evaluate your cardiovascular and bone health are performed. The details and timing of the tests are explained below.

VISIT #1 During the first visit, a research doctor or assistant explains the procedures in detail and answers questions. Blood is drawn (about 1-2 tablespoons) to confirm the diagnosis of hyperparathyroidism and get baseline blood values.

VISIT #2-4 During the following visits, a variety of procedures are performed to evaluate cardiovascular and bone health. The details of the procedures and when they will be performed are outlined below.

1. Blood tests are performed at each visit. Approximately 1-2 tablespoons of blood will be drawn at each visit.
2. A 24-hour urine collection is done 3 times during the 2 year study.
3. Bone mineral density testing (known as DXA) is performed at baseline, 12 and 24 months after enrollment.
4. Carotid Ultrasound: At the baseline visit, 12 and 24 months after enrollment, carotid ultrasound is performed.
5. Echocardiogram: At the baseline visit, 12 and 24 months after enrollment, an echocardiogram is performed.
6. Endothelial Function: At baseline, 6 and 12 months after enrollment, flow mediated dilation of the brachial artery is performed.

ELIGIBILITY:
Inclusion Criteria:

-Primary Hyperparathyroidism

Exclusion Criteria:

* Current use of oral bisphosphonates
* Addition or change in cholesterol lowering medication
* impaired renal function (creatinine >2.0 mg/dl)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults age 50 to 75 with Primary Hyperparathyroidism
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2005-10; Primary Completion 2009-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Structural evidence of increased vascular stiffness or cardiovascular calcification in patients with mild asymptomatic PHPT | 2 years
  To determine whether or not there is structural evidence of increased vascular stiffness or cardiovascular calcification in patients with mild asymptomatic PHPT as compared to matched healthy controls, and to determine the reversibility of these manifestations after successful parathyroidectomy

SECONDARY OUTCOMES:
Evidence of abnormal cardiovascular function in patients with mild asymptomatic PHPT | 2 years
  To determine whether or not there is evidence of abnormal cardiovascular function in patients with mild asymptomatic PHPT, and to determine the reversibility of these manifestations after successful parathyroidectomy
Evidence of abnormal cardiovascular structure or function in patients with asymptomatic PHPT who meet NIH Guidelines for Surgery | 2 years
  To determine whether or not there is evidence of abnormal cardiovascular structure or function in patients with asymptomatic PHPT who meet NIH Guidelines for Surgery, and to determine the reversibility of these manifestations after successful parathyroidectomy

OTHER OUTCOMES:
To determine the association between the severity of PHPT and the presence of altered cardiovascular structure and function | 2 years
  To determine the association between the severity of PHPT and the presence of altered cardiovascular structure and function as assessed in outcomes 1 to 3

CONTACTS AND LOCATIONS:
Overall Officials: Shonni J Silverberg, MD, Principal Investigator — Columbia University
Locations (1):
- Metabolic Bone Diseases Unit, New York, New York, United States

REFERENCES:
- [Derived] Camporese G, Bernardi E, Bortoluzzi C, Noventa F, Hong NV, Callegari E, Villalta S, Tonello C, Nardin M, Campello E, Spiezia L, Simioni P. MAC Project-Monitoring Anticoagulant Therapy Observational Study: Rationale and Protocol. Front Med (Lausanne). 2021 Jan 28;7:584459. doi: 10.3389/fmed.2020.584459. eCollection 2020. PMID 33585500